CLINICAL TRIAL: NCT01777698
Title: Body Composition Analysis by Bioelectrical Impedance Vector Analysis in Patients With Hepatocellular Carcinoma Undergoing Chemoembolization.
Brief Title: Body Composition Analysis in Patients Undergoing Chemoembolization
Status: Completed | Type: Observational
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Principal Investigator, ALDO TORRE DELGADILLO, M.D., M.Sc., Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Other Study IDs: QMECR1
Record Dates: First submitted 2013-01-21; First posted 2013-01-29 (Estimated); Last update posted 2016-06-08 (Estimated); Status verified 2016-06

CONDITIONS: Hepatocellular Carcinoma
Keywords: body composition; hepatocellular carcinoma; chemoembolization
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Hepatocellular carcinoma represents 80-90% of primary hepatic malignant tumors. 80% of patients with hepatocellular carcinoma are associated with cirrhosis.

Chemoembolization is a process in which a chemotherapeutic agent is deposited directly into the hepatic tumor where the principal artery is embolized.

Bioelectrical impedance bases its evaluation in a model where the body is conformed by two different compartments: fat mass and fat free mass.

Bioelectrical impedance is complemented by vectorial analysis, which is independent to the state of hydration and is helpful to monitor any changes in corporal composition. It can be used as a control for the interpretation of the bioelectrical impedance.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hepato-renal disease
* Patients with hepatocellular carcinoma that are put down to radiofrequency ablation
* Patients with depression or any psiquiatric disease.
* Patients that don't agree to participate in the project.

Exclusion Criteria:

* Patients with hepatocellular carcinoma that are put down to radiofrequency ablation
* Patients with depression or any psiquiatric disease.
* Patients that don't agree to participate in the project.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients will be recruited from the Radiology Department of a tertiary care center.
Sampling Method: Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2012-04; Primary Completion 2015-08 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Changes in body composition | 1 hour before treatment, 2 weeks after treatment, and 1 month after treatment
  To evaluate any changes in corporal composition in patients undergoing chemoembolization.

CONTACTS AND LOCATIONS:
Overall Officials: Aldo Torre, M.D, M.Sc., Study Chair — Instituto Nacional de Nutrición y Ciencias Médicas "Salvador Zubirán"
Locations (1):
- Instituto Nacional de Ciencias Médicas y Nutrición "Salvador Zubirán", Mexico City, Mexico